CLINICAL TRIAL: NCT02349425
Title: A Dose Escalation Study to Assess the Efficacy and Tolerance of AF-219 in Subjects With Refractory Chronic Cough
Brief Title: A Dose Escalation Study of Gefapixant (AF-219/MK-7264) in Refractory Chronic Cough (MK-7264-010)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7264-010; AF219-010 (Other: Afferent Pharmaceuticals); MK-7264-010 (Other: Merck Protocol Number); 2015-000474-35 (Other: EudraCT Number)
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Gefapixant>Placebo (Experimental): 50, 100, 150, and 200 mg gefapixant twice daily (BID) for 4 days each in Period 1 and placebo BID for 16 days in Period 2. For Cohort 1, there was a 3 to 7 day washout period between treatment periods.
  Interventions: Drug: Gefapixant; Drug: Placebo (for gefapixant)
- Cohort 1: Placebo>Gefapixant (Experimental): Placebo BID for 16 days in Period 1 and gefapixant 50, 100, 150, and 200 mg BID for 4 days each in Period 2. For Cohort 1, there was a 3 to 7 day washout period between treatment periods.
  Interventions: Drug: Gefapixant; Drug: Placebo (for gefapixant)
- Cohort 2: Gefapixant>Placebo (Experimental): Gefapixant 7.5, 15, 30, and 50 mg BID for 4 days each in Period 1 and placebo BID for 16 days in Period 2. For Cohort 2, there was a 14 to 21 day washout period between treatment periods.
  Interventions: Drug: Gefapixant; Drug: Placebo (for gefapixant)
- Cohort 2: Placebo>Gefapixant (Experimental): Placebo BID for 16 days in Period 1 and gefapixant 7.5, 15, 30, and 50 mg BID for 4 days each in Period 2. For Cohort 2, there was a 14 to 21 day washout period between treatment periods.
  Interventions: Drug: Gefapixant; Drug: Placebo (for gefapixant)

INTERVENTIONS:
Drug: Gefapixant — Gefapixant 7.5 and 50mg tablets administered orally
  Other Names: AF-219; MK-7264
Drug: Placebo (for gefapixant) — Placebo to gefapixant 7.5 and 50mg tablets administered orally

SUMMARY:
A randomized, double-blind, placebo-controlled, crossover, dose escalation study to assess the efficacy and tolerability of gefapixant (AF-219; MK-7264) in participants with refractory chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiograph or computed tomography (CT) thorax within the last 12 months not demonstrating any abnormality considered to be significantly contributing to the chronic cough
* Refractory chronic cough for at least one year: a cough that is unresponsive to at least 8 weeks of targeted treatment for identified underlying triggers including reflux disease, asthma and post-nasal drip or unexplained cough: a cough for which no objective evidence of an underlying trigger can be determined after investigation
* Score of ≥ 40 mm on the Cough Severity Visual Analog Scale (VAS) at Screening
* Women of child-bearing potential must use 2 forms of acceptable birth control method from Screening through the Follow-Up Visit.
* Male participants and their partners of child-bearing potential must use 2 methods of acceptable birth control from Screening until 3 months after the last dose of study drug.
* Written informed consent.
* Willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

* Current smoker
* Individuals who have given up smoking within the past 6 months, or those with >20 pack-year smoking history
* Treatment with an angiotensin converting enzyme (ACE)-inhibitor as the potential cause of a participant's cough, or requiring treatment with an ACE-inhibitor during the study or within 4 weeks prior to the Baseline Visit (Day 0)
* Forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 60%
* History of upper respiratory tract infection or recent significant change in pulmonary status within 4 weeks of the Baseline Visit (Day 0)
* History of opioid use within 1 week of the Baseline Visit (Day 0)
* Requiring concomitant therapy with prohibited medications
* Body mass index (BMI) <18 kg/m^2 or ≥ 37 kg/m^2
* History of concurrent malignancy or recurrence of malignancy within 2 years prior to Screening (not including participants with <3 excised basal cell carcinomas)
* History of a diagnosis of drug or alcohol dependency or abuse within approximately the last 3 years
* Any condition possibly affecting drug absorption (e.g., gastrectomy, gastroplasty, any type of bariatric surgery, vagotomy, or bowel resection)
* Screening systolic blood pressure (SBP) >160 mmHg or a diastolic blood pressure (DBP) >90 mmHg
* Clinically significant abnormal electrocardiogram (ECG) at Screening
* Personal or family history of congenital long QT syndrome or family history of sudden death
* Cardiac pacemaker
* Significantly abnormal laboratory tests at Screening
* Breastfeeding
* Treatment with an investigational drug (except gefapixant) or biologic within 60 days preceding the first dose of study medication or plans to take another investigational drug or biologic within 30 days of study completion
* Blood donation within 56 days or plasma donation within 7 days prior to dosing
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Smith JA, Kitt MM, Butera P, Smith SA, Li Y, Xu ZJ, Holt K, Sen S, Sher MR, Ford AP. Gefapixant in two randomised dose-escalation studies in chronic cough. Eur Respir J. 2020 Mar 20;55(3):1901615. doi: 10.1183/13993003.01615-2019. Print 2020 Mar. PMID 31949115
- See also: P2X3 Receptor Antagonist (AF-219) in Refractory Chronic Cough: A Randomised, Double-Blind, Placebo-Controlled Phase 2 Study — http://dx.doi.org/10.1016/S0140-6736(14)61255-1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 12 clinical trial sites in the United States.
Pre-assignment Details: 29 participants were enrolled, randomized and treated with study drug in Cohort 1 and 30 participants in Cohort 2. Of the 30 participants in Cohort 2, 18 of them were from Cohort 1 and they re-consented, were given new randomization numbers and treated with study drug.
Groups:
- Cohort 1: Gefapixant>Placebo: Gefapixant 50, 100, 150, and 200 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 1 and placebo to gefapixant 50, 100, 150, and 200 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 2. For Cohort 1, there was a 3 to 7 day washout period between treatment periods.
- Cohort 1: Placebo>Gefapixant: Placebo to gefapixant 50, 100, 150, and 200 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 1 and gefapixant 50, 100, 150, and 200 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 2. For Cohort 1, there was a 3 to 7 day washout period between treatment periods.
- Cohort 2: Gefapixant>Placebo: Gefapixant 7.5, 15, 30, and 50 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 1 and placebo to gefapixant 7.5, 15, 30, and 50 mg, tablet(s) administered by mouth twice daily for 4 days each in Period 2. For Cohort 2 there was a 14-21 day washout period between treatment periods.
- Cohort 2: Placebo>Gefapixant: Placebo to gefapixant 7.5, 15, 30, and 50 mg, tablet(s) administered by mouth twice daily for 4 days each in Period 1 and gefapixant 7.5, 15, 30, and 50 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 2. For Cohort 2 there was a 14-21 day washout period between treatment periods.
Period: Period 1
Arm/Group | Cohort 1: Gefapixant>Placebo | Cohort 1: Placebo>Gefapixant | Cohort 2: Gefapixant>Placebo | Cohort 2: Placebo>Gefapixant
Started | 15 | 14 | 15 | 15
Completed | 14 | 13 | 15 | 15
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Period: Period 2
Arm/Group | Cohort 1: Gefapixant>Placebo | Cohort 1: Placebo>Gefapixant | Cohort 2: Gefapixant>Placebo | Cohort 2: Placebo>Gefapixant
Started | 14 | 13 | 15 | 15
Completed | 14 | 12 | 14 | 15
Not Completed | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all randomized participants who have received at least 1 dose of study drug.
Groups:
- Cohort 1 - Gefapixant>Placebo: Gefapixant 50, 100, 150, and 200 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 1 and placebo to gefapixant 50, 100, 150, and 200 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 2. For Cohort 1, there was a 3 to 7-day washout period between treatment periods.
- Cohort 1 - Placebo>Gefalixant: Placebo to gefapixant 50, 100, 150, and 200 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 1 and gefapixant 50, 100, 150, and 200 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 2. For Cohort 1, there was a 3 to 7 day washout period between treatment periods.
- Cohort 2 - Gefapixant>Placebo: Gefapixant 7.5, 15, 30 and 50 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 1 and placebo to gefapixant 7.5, 15, 30 and 50 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 2. For Cohort 2, there was a 14 to 21-day washout period between treatment periods.
- Cohort 2 - Placebo>Gefapixant: Placebo to gefapixant 7.5, 15, 30 and 50 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 1 and gefapixant 7.5, 15, 30 and 50 mg, tablet(s) administered by mouth, twice daily, for 4 days each in Period 2. For Cohort 2, there was a 14 to 21-day washout period between treatment periods.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Gefapixant>Placebo | Cohort 1 - Placebo>Gefalixant | Cohort 2 - Gefapixant>Placebo | Cohort 2 - Placebo>Gefapixant | Total
Number analyzed (Participants) | 15 | 14 | 15 | 15 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (6.92) | 61.7 (7.77) | 60.7 (9.42) | 59.8 (12.8) | 61.7 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 12 | 12 | 49
  Male | 2 | 2 | 3 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 14 | 14 | 14 | 14 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 15 | 13 | 13 | 15 | 56
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Awake Objective Cough Frequency on Log-transformed Scale - Cohort 1
Description: Awake Objective Frequency (per hour) is the total number of cough events during the monitoring period (in general, 24-hr interval) the participant is awake divided by the total duration (in hours) for the monitoring period the participant is awake. 24-hour sound recordings were collected using a digital recording device.
Time Frame: Period 1 (while awake): baseline (Day 0) and 24 hours after Day 4, 8, 12 & 16 doses; Period 2 (while awake): baseline (Day 22) and 24 hours after Day 26, 30, 34 and 38 doses
Population: Analysis population consisted of all participants in Cohort 1 for Periods 1 and 2 who were randomized, received at least 1 dose of study drug, were compliant with the study procedure and had available data for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Log coughs/hour
Groups:
- Cohort 1 - Gefapixant 50 mg: Gefapixant 50 mg tablet administered by mouth BID for 4 days.
- Cohort 1 - Placebo for Gefapixant 50 mg; Cohort 1 - Placebo for Gefapixant 100 mg; Cohort 1 - Placebo for Gefapixant 150 mg; Cohort 1 - Placebo for Gefapixant 200 mg: Placebo tablet administered by mouth BID for 4 days.
- Cohort 1 - Gefapixant 100 mg: Gefapixant 100 mg tablet administered by mouth BID for 4 days.
- Cohort 1 - Gefapixant 150 mg: Gefapixant 150 mg tablet administered by mouth BID for 4 days.
- Cohort 1 - Gefapixant 200 mg: Gefapixant 200 mg tablet administered by mouth BID for 4 days.
Arm/Group | Cohort 1 - Gefapixant 50 mg | Cohort 1 - Placebo for Gefapixant 50 mg | Cohort 1 - Gefapixant 100 mg | Cohort 1 - Placebo for Gefapixant 100 mg | Cohort 1 - Gefapixant 150 mg | Cohort 1 - Placebo for Gefapixant 150 mg | Cohort 1 - Gefapixant 200 mg | Cohort 1 - Placebo for Gefapixant 200 mg
Number analyzed (Participants) | 26 | 25 | 24 | 25 | 23 | 22 | 25 | 25
Log coughs/hour | 0.56 [0.43 to 0.72] | 0.95 [0.73 to 1.23] | 0.46 [0.34 to 0.61] | 0.95 [0.71 to 1.28] | 0.48 [0.35 to 0.65] | 0.90 [0.65 to 1.24] | 0.45 [0.33 to 0.63] | 1.06 [0.75 to 1.48]
Statistical Analysis 1: Comparison: Cohort 1 - Gefapixant 50 mg vs Cohort 1 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.0055, Mixed Models Analysis; Per protocol, statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -41.222, 95% CI 2-sided [-59.294 to -15.127] — Percent change difference between Gefapixant and placebo was estimated by 100 x [e^diff - 1] where e=exponent of difference; and diff = the treatment mean difference from mixed model of change from baseline based on log-transformed data
Statistical Analysis 2: Comparison: Cohort 1 - Gefapixant 100 mg vs Cohort 1 - Placebo for Gefapixant 100 mg; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Per protocol, statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -51.973, 95% CI 2-sided [-68.230 to -27.397] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort 1 - Gefapixant 150 mg vs Cohort 1 - Placebo for Gefapixant 150 mg; Test type: Superiority; p = 0.0075, Mixed Models Analysis; Per protocol, statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -46.853, 95% CI 2-sided [-66.291 to -16.206] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort 1 - Gefapixant 200 mg vs Cohort 1 - Placebo for Gefapixant 200 mg; Test type: Superiority; p = 0.0009, Mixed Models Analysis; Per protocol, statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -57.067, 95% CI 2-sided [-73.375 to -30.771] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change in Awake Objective Cough Frequency on Log-transformed Scale - Cohort 2
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Analysis population consisted of all participants in Cohort 2 for Periods 1 and 2 who were randomized, received at least 1 dose of study drug, were compliant with the study procedure and had available data for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Log coughs/hour
Groups:
- Cohort 2 - Gefapixant 7.5 mg: Gefapixant 7.5 mg tablet administered by mouth BID for 4 days.
- Cohort 2 - Placebo for Gefapixant 7.5 mg; Cohort 2 - Placebo for Gefapixant 15 mg; Cohort 2 - Placebo for Gefapixant 30 mg; Cohort 2 - Placebo for Gefapixant 50 mg: Placebo tablet administered by mouth BID for 4 days.
- Cohort 2 - Gefapixant 15 mg: Gefapixant 15 mg tablet administered by mouth BID for 4 days.
- Cohort 2 - Gefapixant 30 mg: Gefapixant 30 mg tablet administered by mouth BID for 4 days.
- Cohort 2 - Gefapixant 50 mg: Gefapixant 50 mg tablet administered by mouth BID for 4 days.
Arm/Group | Cohort 2 - Gefapixant 7.5 mg | Cohort 2 - Placebo for Gefapixant 7.5 mg | Cohort 2 - Gefapixant 15 mg | Cohort 2 - Placebo for Gefapixant 15 mg | Cohort 2 - Gefapixant 30 mg | Cohort 2 - Placebo for Gefapixant 30 mg | Cohort 2 - Gefapixant 50 mg | Cohort 2 - Placebo for Gefapixant 50 mg
Number analyzed (Participants) | 29 | 28 | 30 | 29 | 29 | 29 | 29 | 27
Log coughs/hour | 0.80 [0.66 to 0.96] | 0.93 [0.77 to 1.13] | 0.67 [0.57 to 0.80] | 0.90 [0.75 to 1.08] | 0.53 [0.40 to 0.69] | 0.84 [0.64 to 1.10] | 0.44 [0.32 to 0.60] | 1.00 [0.72 to 1.38]
Statistical Analysis 1: Comparison: Cohort 2 - Gefapixant 7.5 mg vs Cohort 2 - Placebo for Gefapixant 7.5 mg; Test type: Superiority; p = 0.2542, Mixed Models Analysis; Per protocol, statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -14.691, 95% CI 2-sided [-35.307 to 12.493] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 2 - Gefapixant 15 mg vs Cohort 2 - Placebo for Gefapixant 15 mg; Test type: Superiority; p = 0.0267, Mixed Models Analysis; Per protocol, statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -25.165, 95% CI 2-sided [-42.014 to -3.4210] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Cohort 2 - Gefapixant 30 mg vs Cohort 2 - Placebo for Gefapixant 30 mg; Test type: Superiority; p = 0.0198, Mixed Models Analysis; Per protocol, statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -37.146, 95% CI 2-sided [-57.345 to -7.3821] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Cohort 2 - Gefapixant 50 mg vs Cohort 2 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.0006, Mixed Models Analysis; Per protocol, statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -55.920, 95% CI 2-sided [-71.923 to -30.797] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Percent Change From Baseline in Awake Cough Frequency for Cohort 1
Description: Awake Objective Cough Frequency (per hour) is the total number of cough events during the monitoring period (in general, 24-hr interval) the participant is awake divided by the total duration (in hours) for the monitoring period the participant is awake. 24-hour sound recordings were collected using a digital recording device. Percent Change in Awake Cough Frequency is the change from baseline in awake cough frequency x 100, divided by baseline awake cough frequency. A negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Cohort 1' - Placebo for Gefapixant 50 mg; Cohort 1 - Placebo for Gefapixant 100 mg; Cohort 1 - Placebo for Gefapixant 150 mg; Cohort 1 - Placebo for Gefapixant 200 mg: Placebo tablet administered by mouth BID for 4 days.
Arm/Group | Cohort 1 - Gefapixant 50 mg | Cohort 1' - Placebo for Gefapixant 50 mg | Cohort 1 - Gefapixant 100 mg | Cohort 1 - Placebo for Gefapixant 100 mg | Cohort 1 - Gefapixant 150 mg | Cohort 1 - Placebo for Gefapixant 150 mg | Cohort 1 - Gefapixant 200 mg | Cohort 1 - Placebo for Gefapixant 200 mg
Number analyzed (Participants) | 26 | 25 | 24 | 25 | 23 | 22 | 25 | 25
Percent Change | -20.6 (84.29) | -0.1 (33.75) | -31.7 (70.27) | 1.9 (35.18) | -22.0 (82.84) | -0.1 (39.55) | -27.9 (57.03) | 15.1 (48.38)

4. Primary Outcome: Percent Change From Baseline in Awake Cough Frequency for Cohort 2
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Cohort 2 - Placebo for Gefapixant 50 mg: Placebo tablets administered by mouth BID for 4 days.
Arm/Group | Cohort 2 - Gefapixant 7.5 mg | Cohort 2 - Placebo for Gefapixant 7.5 mg | Cohort 2 - Gefapixant 15 mg | Cohort 2 - Placebo for Gefapixant 15 mg | Cohort 2 - Gefapixant 30 mg | Cohort 2 - Placebo for Gefapixant 30 mg | Cohort 2 - Gefapixant 50 mg | Cohort 2 - Placebo for Gefapixant 50 mg
Number analyzed (Participants) | 29 | 28 | 30 | 29 | 29 | 29 | 29 | 27
Percent Change | 5.0 (125.05) | -3.8 (36.13) | -21.4 (39.32) | -6.4 (33.78) | -26.3 (61.01) | -1.1 (64.38) | -28.1 (74.90) | 23.1 (92.60)

5. Primary Outcome: Responder Analysis of Awake Cough Frequency for Cohort 1
Description: Participants were classified as responders based on the magnitude of the percent change from baseline in Awake Objective cough frequency: 1. ≥70% Reduction=1 if Percent Change from Baseline in cough frequency at the end of the dosing interval ≤-70.0%; 0 Otherwise; 2. ≥50% Reduction=1 if Percent Change from Baseline in cough frequency at the end of the dosing interval ≤ -50.0%; 0 Otherwise; 3. ≥30% Reduction=1 if Percent Change from Baseline in cough frequency at the end of the dosing interval ≤ -30.0%; 0 Otherwise. These responder definitions were not mutually exclusive. A participant who achieved a 1 for ≥70% Reduction for a particular period and dosing interval, were by definition, classified as ≥50% Reduction and ≥ 30% Reduction.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percent Responders
Arm/Group | Cohort 1 - Gefapixant 50 mg | Cohort 1 - Placebo for Gefapixant 50 mg | Cohort 1 - Gefapixant 100 mg | Cohort 1 - Placebo for Gefapixant 100 mg | Cohort 1 - Gefapixant 150 mg | Cohort 1 - Placebo for Gefapixant 150 mg | Cohort 1 - Gefapixant 200 mg | Cohort 1 - Placebo for Gefapixant 200 mg
Number analyzed (Participants) | 26 | 25 | 24 | 25 | 23 | 22 | 25 | 25
Percent Responders
  % Reduction ≥70 | 34.6 | 0 | 33.3 | 0 | 34.8 | 4.5 | 32.0 | 0
  % Reduction ≥50 | 46.2 | 0 | 50.0 | 4.0 | 47.8 | 4.5 | 44.0 | 0
  % Reduction ≥30 | 53.8 | 12.0 | 66.7 | 16.0 | 65.2 | 22.7 | 56.0 | 16.0

6. Primary Outcome: Responder Analysis of Awake Cough Frequency for Cohort 2
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: Percent Responders
Arm/Group | Cohort 2 - Gefapixant 7.5 mg | Cohort 2 - Placebo for Gefapixant 7.5 mg | Cohort 2 - Gefapixant 15 mg | Cohort 2 - Placebo for Gefapixant 15 mg | Cohort 2 - Gefapixant 30 mg | Cohort 2 - Placebo for Gefapixant 30 mg | Cohort 2 - Gefapixant 50 mg | Cohort 2 - Placebo for Gefapixant 50 mg
Number analyzed (Participants) | 29 | 28 | 30 | 29 | 29 | 29 | 29 | 27
Percent Responders
  % Reduction ≥70 | 3.4 | 3.6 | 10.0 | 0 | 20.7 | 3.4 | 31.0 | 3.7
  % Reduction ≥50 | 13.8 | 7.1 | 20.0 | 6.9 | 31.0 | 17.2 | 41.4 | 11.1
  % Reduction ≥30 | 37.9 | 14.3 | 46.7 | 20.7 | 62.1 | 31.0 | 55.2 | 22.2

7. Secondary Outcome: Change From Baseline in Awake (0-8 Hours) Objective Cough Frequency for Cohort 1
Description: Awake (0-8 hours) Objective Cough Frequency is the total number of cough events during the monitoring period the participant was awake for the first 8 hours after the participant took their study medication divided by 8 or the total duration (in hours) for the monitoring period the participant was awake whichever is less. 24-hour sound recordings were collected using a digital recording device. Results are change from baseline: a negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency.
  Cough frequency was analyzed using a mixed model repeated measures (MMRM) to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Period 1 (while awake): baseline (Day 0) and 0-8 hours after Day 4, 8, 12 & 16 doses; Period 2 (while awake): baseline (Day 22) and 0-8 hours after Day 26, 30, 34 and 38 doses
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Cohort 1 - Gefapixant 50 mg | Cohort 1 - Placebo for Gefapixant 50 mg | Cohort 1 - Gefapixant 100 mg | Cohort 1 - Placebo for Gefapixant 100 mg | Cohort 1 - Gefapixant 150 mg | Cohort 1 - Placebo for Gefapixant 150 mg | Cohort 1 - Gefapixant 200 mg | Cohort 1 - Placebo for Gefapixant 200 mg
Number analyzed (Participants) | 26 | 25 | 24 | 25 | 23 | 22 | 25 | 25
Coughs/hour | -24.5 [-33.0 to -15.9] | -5.5 [-14.2 to 3.3] | -24.5 [-33.1 to -15.8] | -0.1 [-8.8 to 8.7] | -26.5 [-40.3 to -12.8] | 2.7 [-11.4 to 16.9] | -27.5 [-37.9 to -17.0] | 2.2 [-8.5 to 12.8]
Statistical Analysis 1: Comparison: Cohort 1 - Gefapixant 50 mg vs Cohort 1 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.003, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -19.0, 95% CI 2-sided [-31.2 to -6.8]
Statistical Analysis 2: Comparison: Cohort 1 - Gefapixant 100 mg vs Cohort 1 - Placebo for Gefapixant 100 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -24.4, 95% CI 2-sided [-36.7 to -12.1]
Statistical Analysis 3: Comparison: Cohort 1 - Gefapixant 150 mg vs Cohort 1 - Placebo for Gefapixant 150 mg; Test type: Superiority; p = 0.005, Mixed Models Analysis; Per protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -29.3, 95% CI 2-sided [-49.0 to -9.5]
Statistical Analysis 4: Comparison: Cohort 1 - Gefapixant 200 mg vs Cohort 1 - Placebo for Gefapixant 200 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -29.6, 95% CI 2-sided [-44.6 to -14.7]

8. Secondary Outcome: Change From Baseline in Awake (0-8 Hours) Objective Cough Frequency for Cohort 2
Description: as for outcome 7
Time Frame: as for outcome 7
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Cohort 2 - Gefapixant 7.5 mg | Cohort 2 - Placebo for Gefapixant 7.5 mg | Cohort 2 - Gefapixant 15 mg | Cohort 2 - Placebo for Gefapixant 15 mg | Cohort 2 - Gefapixant 30 mg | Cohort 2 - Placebo for Gefapixant 30 mg | Cohort 2 - Gefapixant 50 mg | Cohort 2 - Placebo for Gefapixant 50 mg
Number analyzed (Participants) | 29 | 28 | 30 | 29 | 29 | 29 | 29 | 27
Coughs/hour | -8.0 [-17.9 to 1.9] | -1.1 [-11.1 to 9.0] | -15.2 [-22.1 to -8.3] | -1.7 [-8.8 to 5.3] | -21.7 [-31.9 to -11.5] | 8.5 [-1.8 to 18.8] | -21.9 [-32.8 to -11.0] | 4.7 [-6.5 to 16.0]
Statistical Analysis 1: Comparison: Cohort 2 - Gefapixant 7.5 mg vs Cohort 2 - Placebo for Gefapixant 7.5 mg; Test type: Superiority; p = 0.332, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -6.9, 95% CI 2-sided [-21.0 to 7.2]
Statistical Analysis 2: Comparison: Cohort 2 - Gefapixant 15 mg vs Cohort 2 - Placebo for Gefapixant 15 mg; Test type: Superiority; p = 0.008, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -13.5, 95% CI 2-sided [-23.3 to -3.6]
Statistical Analysis 3: Comparison: Cohort 2 - Gefapixant 30 mg vs Cohort 2 - Placebo for Gefapixant 30 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -30.2, 95% CI 2-sided [-44.7 to -15.7]
Statistical Analysis 4: Comparison: Cohort 2 - Gefapixant 50 mg vs Cohort 2 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -26.7, 95% CI 2-sided [-42.3 to -11.0]

9. Secondary Outcome: Change From Baseline in Total (24 Hours) Cough Frequency - Cohort 1
Description: Total (0-24 hours) Objective Cough Frequency is the total number of cough events during the monitoring period divided by the total duration (in hours, i.e., 24 hours mostly) for the monitoring period. 24-hour sound recordings were collected using a digital recording device. Results are change from baseline: a negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency.
  Cough frequency was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Period 1: baseline (Day 0) and 0-24 hours after Day 4, 8, 12 & 16 doses; Period 2: baseline (Day 22) and 0-24 hours after Day 26, 30, 34 and 38 doses
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Cohort 1 - Gefapixant 50 mg | Cohort 1 - Placebo for Gefapixant 50 mg | Cohort 1 - Gefapixant 100 mg | Cohort 1 - Placebo for Gefapixant 100 mg | Cohort 1 - Gefapixant 150 mg | Cohort 1 - Placebo for Gefapixant 150 mg | Cohort 1 - Gefapixant 200 mg | Cohort 1 - Placebo for Gefapixant 200 mg
Number analyzed (Participants) | 26 | 25 | 24 | 25 | 23 | 22 | 25 | 25
Coughs/hour | -16.6 [-22.4 to -10.9] | -1.5 [-7.5 to 4.5] | -17.6 [-24.1 to -11.0] | -0.9 [-7.5 to 5.8] | -18.0 [-26.1 to -9.9] | 1.5 [-6.8 to 9.8] | -17.4 [-25.2 to -9.5] | 3.1 [-4.9 to 11.2]
Statistical Analysis 1: Comparison: Cohort 1 - Gefapixant 50 mg vs Cohort 1 - Placebo for Gefapixant 50 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -15.2, 95% CI 2-sided [-23.5 to -6.8]
Statistical Analysis 2: Comparison: Cohort 1 - Gefapixant 100 mg vs Cohort 1 - Placebo for Gefapixant 100 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -16.7, 95% CI 2-sided [-26.1 to -7.4]
Statistical Analysis 3: Comparison: Cohort 1 - Gefapixant 150 mg vs Cohort 1 - Placebo for Gefapixant 150 mg; Test type: Superiority; p = 0.002, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -19.5, 95% CI 2-sided [-31.1 to -7.8]
Statistical Analysis 4: Comparison: Cohort 1 - Gefapixant 200 mg vs Cohort 1 - Placebo for Gefapixant 200 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -20.5, 95% CI 2-sided [-31.8 to -9.3]

10. Secondary Outcome: Change From Baseline in Total (24 Hours) Cough Frequency - Cohort 2
Description: as for outcome 9
Time Frame: as for outcome 9
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Cohort 2 - Gefapixant 7.5 mg | Cohort 2 - Placebo for Gefapixant 7.5 mg | Cohort 2 - Gefapixant 15 mg | Cohort 2 - Placebo for Gefapixant 15 mg | Cohort 2 - Gefapixant 30 mg | Cohort 2 - Placebo for Gefapixant 30 mg | Cohort 2 - Gefapixant 50 mg | Cohort 2 - Placebo for Gefapixant 50 mg
Number analyzed (Participants) | 29 | 28 | 30 | 29 | 29 | 29 | 29 | 27
Coughs/hour | -6.9 [-12.6 to -1.1] | -2.7 [-8.6 to 3.1] | -11.0 [-15.5 to -6.4] | -3.8 [-8.4 to 0.9] | -16.9 [-23.3 to -10.4] | 1.4 [-5.2 to 7.9] | -15.9 [-21.0 to -9.9] | 1.8 [-4.4 to 7.9]
Statistical Analysis 1: Comparison: Cohort 2 - Gefapixant 7.5 mg vs Cohort 2 - Placebo for Gefapixant 7.5 mg; Test type: Superiority; p = 0.315, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-12.3 to 4.0]
Statistical Analysis 2: Comparison: Cohort 2 - Gefapixant 15 mg vs Cohort 2 - Placebo for Gefapixant 15 mg; Test type: Superiority; p = 0.030, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-13.7 to -0.7]
Statistical Analysis 3: Comparison: Cohort 2 - Gefapixant 30 mg vs Cohort 2 - Placebo for Gefapixant 30 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -18.2, 95% CI 2-sided [-27.4 to -9.1]
Statistical Analysis 4: Comparison: Cohort 2 - Gefapixant 50 mg vs Cohort 2 - Placebo for Gefapixant 50 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -17.6, 95% CI 2-sided [-26.3 to -9.0]

11. Secondary Outcome: Change From Baseline in Sleep Cough Frequency - Cohort 1
Description: Sleep Objective Cough Frequency is the total number of cough events during the monitoring period the participant is asleep divided by the total duration (in hours) for the monitoring period the participant is asleep. 24-hour sound recording were collected with a digital recording device. Results are change from baseline: a negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency.
  Cough frequency was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Period 1 (while asleep): baseline (Day 0) and 24 hours after Day 4, 8, 12 & 16 doses; Period 2 (while asleep): baseline (Day 22) and 24 hours after Day 26, 30, 34 and 38 doses
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Coughs/hour
Arm/Group | Cohort 1 - Gefapixant 50 mg | Cohort 1 - Placebo for Gefapixant 50 mg | Cohort 1 - Gefapixant 100 mg | Cohort 1 - Placebo for Gefapixant 100 mg | Cohort 1 - Gefapixant 150 mg | Cohort 1 - Placebo for Gefapixant 150 mg | Cohort 1 - Gefapixant 200 mg | Cohort 1 - Placebo for Gefapixant 200 mg
Number analyzed (Participants) | 24 | 24 | 21 | 24 | 22 | 22 | 24 | 25
Coughs/hour | -3.5 [-7.0 to 0.1] | 0.1 [-3.5 to 3.7] | -3.1 [-6.8 to 0.6] | -0.7 [-4.2 to 2.8] | -2.0 [-4.8 to 0.7] | -0.1 [-2.8 to 2.6] | -3.6 [-7.0 to -0.1] | 0.2 [-3.2 to 3.6]
Statistical Analysis 1: Comparison: Cohort 1 - Gefapixant 50 mg vs Cohort 1 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.169, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-8.6 to 1.6]
Statistical Analysis 2: Comparison: Cohort 1 - Gefapixant 100 mg vs Cohort 1 - Placebo for Gefapixant 100 mg; Test type: Superiority; p = 0.341, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-7.5 to 2.6]
Statistical Analysis 3: Comparison: Cohort 1 - Gefapixant 150 mg vs Cohort 1 - Placebo for Gefapixant 150 mg; Test type: Superiority; p = 0.311, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-5.8 to 1.9]
Statistical Analysis 4: Comparison: Cohort 1 - Gefapixant 200 mg vs Cohort 1 - Placebo for Gefapixant 200 mg; Test type: Superiority; p = 0.128, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-8.6 to 1.1]

12. Secondary Outcome: Change From Baseline in Sleep Cough Frequency - Cohort 2
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Coughs/hour
Groups:
- Cohort 2 - Placebo for Gefapixant 7.5 mg: Placebo tablet administered by mouth BID for 4 days. .
Arm/Group | Cohort 2 - Gefapixant 7.5 mg | Cohort 2 - Placebo for Gefapixant 7.5 mg | Cohort 2 - Gefapixant 15 mg | Cohort 2 - Placebo for Gefapixant 15 mg | Cohort 2 - Gefapixant 30 mg | Cohort 2 - Placebo for Gefapixant 30 mg | Cohort 2 - Gefapixant 50 mg | Cohort 2 - Placebo for Gefapixant 50 mg
Number analyzed (Participants) | 29 | 28 | 30 | 29 | 29 | 29 | 28 | 27
Coughs/hour | 0.6 [-2.7 to 3.9] | -0.6 [-3.9 to 2.8] | -3.1 [-5.6 to -0.5] | -2.5 [-5.1 to 0.2] | -2.4 [-4.7 to -0.2] | -1.6 [-3.8 to 0.7] | -3.0 [-8.7 to 2.6] | 2.1 [-3.6 to 7.9]
Statistical Analysis 1: Comparison: Cohort 2 - Gefapixant 7.5 mg vs Cohort 2 - Placebo for Gefapixant 7.5 mg; Test type: Superiority; p = 0.613, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-3.5 to 5.9]
Statistical Analysis 2: Comparison: Cohort 2 - Gefapixant 15 mg vs Cohort 2 - Placebo for Gefapixant 15 mg; Test type: Superiority; p = .743, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-4.3 to 3.1]
Statistical Analysis 3: Comparison: Cohort 2 - Gefapixant 30 mg vs Cohort 2 - Placebo for Gefapixant 30 mg; Test type: Superiority; p = 0.589, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-4.1 to 2.3]
Statistical Analysis 4: Comparison: Cohort 2 - Gefapixant 50 mg vs Cohort 2 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.205, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-13.2 to 2.9]

13. Secondary Outcome: Change From Baseline of the Mean Total Daily Cough Severity Diary (CSD) Score for Cohort 1
Description: The daily CSD Score is calculated using the daily CSD instrument, a 7-item, disease specific, patient-reported outcome measure with a recall period of "today" (the current day). The measure evaluates frequency of cough (3 items); intensity of cough (2 items); and sleep disruption due to cough (2 items). Each of these 7 items is rated on an 11-point scale, ranging from 0 (best) to 10 (worst), with higher scores indicating greater severity. The total daily CSD score is the sum of these 7 item scores (Min=0, Max=70). Baseline CSD score = average of CSD scores at screening and baseline. Results are change from baseline: a negative result indicates a decrease in cough severity, while a positive result indicates an increase in cough severity.
  CSD was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Screening; Period 1: baseline (Day 0) and Days 1-17; Period 2: baseline (Day 22) and Days 23-39
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Cohort 1 - Gefapixant 50 mg | Cohort 1 - Placebo for Gefapixant 50 mg | Cohort 1 - Gefapixant 100 mg | Cohort 1 - Placebo for Gefapixant 100 mg | Cohort 1 - Gefapixant 150 mg | Cohort 1 - Placebo for Gefapixant 150 mg | Cohort 1 - Gefapixant 200 mg | Cohort 1 - Placebo for Gefapixant 200 mg
Number analyzed (Participants) | 27 | 27 | 26 | 27 | 26 | 27 | 28 | 28
Score on a scale | -0.6 [-1.2 to -0.1] | 0.0 [-0.5 to 0.5] | -1.1 [-1.8 to -0.5] | 0.1 [-0.5 to 0.8] | -1.5 [-2.2 to -0.8] | 0.1 [-0.6 to 0.8] | -1.6 [-2.4 to -0.8] | 0.1 [-0.7 to 0.9]
Statistical Analysis 1: Comparison: Cohort 1 - Gefapixant 50 mg vs Cohort 1 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.0811, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.4 to 0.1]
Statistical Analysis 2: Comparison: Cohort 1 - Gefapixant 100 mg vs Cohort 1 - Placebo for Gefapixant 100 mg; Test type: Superiority; p = 0.0097, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.2 to -0.3]
Statistical Analysis 3: Comparison: Cohort 1 - Gefapixant 150 mg vs Cohort 1 - Placebo for Gefapixant 150 mg; Test type: Superiority; p = 0.0025, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.6 to -0.6]
Statistical Analysis 4: Comparison: Cohort 1 - Gefapixant 200 mg vs Cohort 1 - Placebo for Gefapixant 200 mg; Test type: Superiority; p = 0.0050, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.8 to -0.5]

14. Secondary Outcome: Change From Baseline of the Mean Total Daily Cough Severity Diary (CSD) Score for Cohort 2
Description: as for outcome 13
Time Frame: Screening; Period 1: baseline (Day 0) and Days 1-17; Period 2: baseline (Day 22) and Days 23-39
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Cohort 1 - Placebo for Gefapixant 15 mg; Cohort 2 - Placebo for Gefapixant 30 mg: Placebo tablet administered by mouth BID for 4 days.
Arm/Group | Cohort 2 - Gefapixant 7.5 mg | Cohort 2 - Placebo for Gefapixant 7.5 mg | Cohort 2 - Gefapixant 15 mg | Cohort 1 - Placebo for Gefapixant 15 mg | Cohort 2 - Gefapixant 30 mg | Cohort 2 - Placebo for Gefapixant 30 mg | Cohort 2 - Gefapixant 50 mg | Cohort 2 - Placebo for Gefapixant 50 mg
Number analyzed (Participants) | 30 | 29 | 30 | 29 | 30 | 29 | 29 | 29
Score on a scale | -1.0 [-1.5 to -0.5] | -0.3 [-0.8 to 0.2] | -1.2 [-1.8 to -0.6] | -0.3 [-0.9 to 0.3] | -1.7 [-2.3 to -1.1] | -0.3 [-1.0 to 0.3] | -1.6 [-2.4 to -0.9] | -0.5 [-1.3 to 0.2]
Statistical Analysis 1: Comparison: Cohort 2 - Gefapixant 7.5 mg vs Cohort 2 - Placebo for Gefapixant 7.5 mg; Test type: Superiority; p = 0.0506, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.4 to 0.0]
Statistical Analysis 2: Comparison: Cohort 2 - Gefapixant 15 mg vs Cohort 1 - Placebo for Gefapixant 15 mg; Test type: Superiority; p = 0.0447, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.7 to -0.0]
Statistical Analysis 3: Comparison: Cohort 2 - Gefapixant 30 mg vs Cohort 2 - Placebo for Gefapixant 30 mg; Test type: Superiority; p = 0.0026, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.2 to -0.5]
Statistical Analysis 4: Comparison: Cohort 2 - Gefapixant 50 mg vs Cohort 2 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.0405, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.2 to -0.0]

15. Secondary Outcome: Change From Baseline at End of Treatment Period Leicester Cough Questionnaire (LCQ): Individual Domain and Total Scores for Cohort 1 and 2
Description: The LCQ-Acute is a 19-item health-related quality-of-life (HRQoL) questionnaire specific for acute cough which contains three domains (i.e., physical, psychological, and social). It is calculated as a mean score for each domain ranging from 1 (worst) to 7 (best), and total score ranging from 3 (worst) to 21 (best). Each item on the LCQ-acute assesses symptoms or the impact of symptoms on HRQoL in the last 24 hours using a 7-point Likert scale ranging from 1 to 7. Higher scores indicate better HRQoL. Participants' perception of their cough severity was assessed, based on the LCQ-Acute score, at Baseline and last day of dose.
  LCQ was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Period 1: Day 0 (baseline) and Day 17; Period 2: Day 22 (baseline) and Day 39
Population: Analysis population consisted of all randomized participants in Periods 1 and 2 who received at least 1 dose of study drug, were compliant with the study procedure and had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Cohort 1 - Gefapixant: Gefapixant 50, 100, 150, and 200 mg tablet(s) administered by mouth BID for 4 days each.
- Cohort 1 - Placebo: Placebo tablet administered by mouth BID for 4 days.
- Cohort 2 - Gefapixant: Gefapixant 7.5, 15, 30, and 50 mg tablet(s) administered by mouth BID for 4 days each.
- Cohort 2 - Placebo: Placebo tablet administered by mouth BID for 4 days each.
Arm/Group | Cohort 1 - Gefapixant | Cohort 1 - Placebo | Cohort 2 - Gefapixant | Cohort 2 - Placebo
Number analyzed (Participants) | 27 | 28 | 30 | 29
Score on a scale | 3.02 [1.61 to 4.42] | -0.82 [-2.19 to 0.55] | 3.57 [2.27 to 4.87] | 0.05 [-1.28 to 1.37]
Statistical Analysis 1: Comparison: Cohort 1 - Gefapixant vs Cohort 1 - Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = 3.84, 95% CI 2-sided [1.88 to 5.80]
Statistical Analysis 2: Comparison: Cohort 2 - Gefapixant vs Cohort 2 - Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = 3.52, 95% CI 2-sided [1.66 to 5.38]

16. Secondary Outcome: Change From Baseline of Cough Visual Analogue Scale (VAS) Score for Cohort 1
Description: Cough VAS is scored from 0 to 100 using a 10 mm visual analogue scale with 0 at 0mm and 100 at 10mm with 0 (no cough) and 100 (most severe cough). Baseline cough VAS is defined as average of screening and baseline cough VAS. Results are change from baseline: a negative result indicates a decrease in cough severity, while a positive result indicates an increase in cough severity.
  Cough VAS was analyzed using MMRM to evaluate the results of the 2-period cross-over study. The derived change measured at each dose were the repeated measures.
Time Frame: Screening; Period 1: baseline (Day 0) and Day 4, 8, 12 & 16; Period 2: baseline (Day 22) and Day 26, 30, 34, 38 and 39
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Cohort 1 - Gefapixant 50 mg | Cohort 1 - Placebo for Gefapixant 50 mg | Cohort 1 - Gefapixant 100 mg | Cohort 1 - Placebo for Gefapixant 100 mg | Cohort 1 - Gefapixant 150 mg | Cohort 1 - Placebo for Gefapixant 150 mg | Cohort 1 - Gefapixant 200 mg | Cohort 1 - Placebo for Gefapixant 200 mg
Number analyzed (Participants) | 27 | 28 | 27 | 27 | 26 | 27 | 26 | 27
Score on a scale | -14.4 [-23.4 to -5.5] | -3.8 [-12.6 to 5.0] | -26.3 [-36.0 to -16.6] | -6.3 [-15.9 to 3.2] | -28.8 [-39.1 to -18.4] | -2.6 [-12.8 to 7.6] | -31.5 [-41.9 to -21.0] | 2.3 [-8.0 to 12.6]
Statistical Analysis 1: Comparison: Cohort 1 - Gefapixant 50 mg vs Cohort 1 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.096, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -10.6, 95% CI 2-sided [-23.2 to 1.9]
Statistical Analysis 2: Comparison: Cohort 1 - Gefapixant 100 mg vs Cohort 1 - Placebo for Gefapixant 100 mg; Test type: Superiority; p = 0.005, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -20.0, 95% CI 2-sided [-33.6 to -6.3]
Statistical Analysis 3: Comparison: Cohort 1 - Gefapixant 150 mg vs Cohort 1 - Placebo for Gefapixant 150 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -26.1, 95% CI 2-sided [-40.7 to -11.6]
Statistical Analysis 4: Comparison: Cohort 1 - Gefapixant 200 mg vs Cohort 1 - Placebo for Gefapixant 200 mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -33.8, 95% CI 2-sided [-48.4 to -19.1]

17. Secondary Outcome: Change From Baseline of Cough Visual Analogue Scale (VAS) Score for Cohort 2
Description: as for outcome 16
Time Frame: Screening; Period 1: baseline (Day 0) and Day 4, 8, 12 & 16; Period 2: baseline (Day 22) and Day 26, 30, 34, 38 and 39
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Cohort 2 - Gefapixant 7.5 mg | Cohort 2 - Placebo for Gefapixant 7.5 mg | Cohort 2 - Gefapixant 15 mg | Cohort 1 - Placebo for Gefapixant 50 mg | Cohort 2 - Gefapixant 30 mg | Cohort 2 - Placebo for Gefapixant 30 mg | Cohort 2 - Gefapixant 50 mg | Cohort 2 - Placebo for Gefapixant 50 mg
Number analyzed (Participants) | 30 | 29 | 30 | 29 | 30 | 29 | 29 | 29
Score on a scale | -12.6 [-21.5 to -3.8] | -6.2 [-15.2 to 2.9] | -17.4 [-26.0 to -8.7] | -10.0 [-18.7 to -1.2] | -23.3 [-31.7 to -14.9] | -7.7 [-16.2 to 0.9] | -24.7 [-35.2 to -14.2] | -9.3 [-19.9 to 1.4]
Statistical Analysis 1: Comparison: Cohort 2 - Gefapixant 7.5 mg vs Cohort 2 - Placebo for Gefapixant 7.5 mg; Test type: Superiority; p = 0.311, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-19.1 to 6.2]
Statistical Analysis 2: Comparison: Cohort 2 - Gefapixant 15 mg vs Cohort 1 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.232, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -7.4, 95% CI 2-sided [-19.7 to 4.9]
Statistical Analysis 3: Comparison: Cohort 2 - Gefapixant 30 mg vs Cohort 2 - Placebo for Gefapixant 30 mg; Test type: Superiority; p = 0.012, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -15.6, 95% CI 2-sided [-27.6 to -3.6]
Statistical Analysis 4: Comparison: Cohort 2 - Gefapixant 50 mg vs Cohort 2 - Placebo for Gefapixant 50 mg; Test type: Superiority; p = 0.043, Mixed Models Analysis; Per Protocol, statistical analysis follows a Mixed Model; Mean Difference (Final Values) = -15.4, 95% CI 2-sided [-30.4 to -0.5]

18. Other Pre Specified Outcome: Baseline (Predose) Awake Objective Cough Frequency for Cohort 1 and Cohort 2
Description: Awake Objective Cough Frequency (per hour) is the total number of cough events during the monitoring period (in general, 24-hr interval) the participant is awake divided by the total duration (in hours) for the monitoring period the participant is awake. 24 hour sound recordings were collected using a digital recording device. Baseline measurements were not available by individual arm because baseline cough frequencies were measured before participants received the first dose of study drug. Baseline summaries were evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: 24 hours (while awake) on Days 0 and 22 (Baseline)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Cohort 1 - Gefapixant | Cohort 1 - Placebo | Cohort 2 - Gefapixant | Cohort 2 - Placebo
Number analyzed (Participants) | 28 | 26 | 30 | 29
Coughs/hour | 54.5 (41.09) | 52.8 (40.44) | 49.6 (44.01) | 46.1 (39.82)

19. Other Pre Specified Outcome: Baseline (Predose) Awake (0 - 8 Hours) Cough Frequency for Cohort 1 and Cohort 2
Description: Awake (0 - 8 hours) Objective Cough Frequency is the total number of cough events during the monitoring period the participant was awake for the first 8 hours after the participant took their study medication divided by 8 or the total duration (in hours) for the monitoring period the participant was awake whichever is less. 24 hour sound recordings were collected with a digital recording device. Baseline measurements were not available by individual arm because baseline cough frequencies were measured before participants received the first dose of study drug. Baseline summaries were evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: First 8 hours (while awake) on Days 0 and 22 (Baseline)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Cohort 1 - Gefapixant | Cohort 1 - Placebo | Cohort 2 - Gefapixant | Cohort 2 - Placebo
Number analyzed (Participants) | 28 | 26 | 30 | 29
Coughs/hour | 51.8 (41.09) | 53.3 (42.30) | 47.2 (42.09) | 42.2 (39.42)

20. Other Pre Specified Outcome: Baseline (Predose) Total (24-hour) Cough Frequency for Cohort 1 and Cohort 2
Description: Total (0 - 24 hours) Objective Cough Frequency is the total number of cough events during the monitoring period divided by the total duration (in hours) for the monitoring period. 24 hour sound recordings were collected using a digital recording device. Baseline measurements were not available by individual arm because baseline cough frequencies were measured before participants received the first dose of study drug. Baseline summaries were evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: 24 hours (while awake) on Days 0 and 22 (Baseline)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Cohort 1 - Gefapixant | Cohort 1 - Placebo | Cohort 2 - Gefapixant | Cohort 2 - Placebo
Number analyzed (Participants) | 28 | 26 | 30 | 29
Coughs/hour | 39.7 (28.38) | 37.9 (27.46) | 36.3 (32.28) | 32.2 (27.97)

21. Other Pre Specified Outcome: Baseline (Predose) for Sleep Cough Frequency for Cohort 1 and Cohort 2
Description: Sleep Objective Cough Frequency is the total number of cough events during the monitoring period the participant is asleep divided by the total duration (in hours) for the monitoring period the participant is asleep. 24-hour sound recording were collected with a digital recording device. Baseline measurements were not available by individual arm because baseline cough frequencies were measured before participants received the first dose of study drug. Baseline summaries were evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: First 8 hours (while asleep) on Days 0 and 22 (Baseline)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Coughs/hour
Arm/Group | Cohort 1 - Gefapixant | Cohort 1 - Placebo | Cohort 2 - Gefapixant | Cohort 2 - Placebo
Number analyzed (Participants) | 27 | 26 | 30 | 29
Coughs/hour | 8.3 (9.30) | 7.8 (9.80) | 10.1 (26.77) | 5.6 (7.58)

22. Other Pre Specified Outcome: Baseline (Predose) for the Mean Total Daily Cough Severity Diary (CSD) Score for Cohort 1 and Cohort 2
Description: The daily CSD Score is calculated using the daily CSD instrument, a 7-item, disease specific, patient-reported outcome measure with a recall period of "today" (the current day). The measure evaluates frequency of cough (3 items); intensity of cough (2 items); and sleep disruption due to cough (2 items). Each of these 7 items is rated on an 11-point scale, ranging from 0 (best) to 10 (worst), with higher scores indicating greater severity. The total daily CSD score is the sum of these 7 item scores (Min=0, Max=70). Baseline CSD score = average of CSD scores at screening and baseline. A negative result indicates a decrease in cough frequency, while a positive result indicates an increase in cough frequency. Baseline measurements were not available by individual arm because baseline cough frequencies were measured before participants received the first dose of study drug. Baseline summaries were evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Baseline (Days 0 and 22)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1 - Gefapixant | Cohort 1 - Placebo | Cohort 2 - Gefapixant | Cohort 2 - Placebo
Number analyzed (Participants) | 28 | 28 | 30 | 28
Score on a scale | 4.2 (1.89) | 3.7 (1.61) | 4.5 (1.98) | 4.5 (1.93)

23. Other Pre Specified Outcome: Baseline (Predose) for the Acute Leicester Cough Questionnaire (LCQ) Instrument for Cohort 1 and Cohort 2
Description: The LCQ-Acute is a 19-item health-related quality-of-life (HRQoL) questionnaire specific for acute cough which contains three domains (i.e., physical, psychological, and social). It is calculated as a mean score for each domain ranging from 1 (worst) to 7 (best), and total score ranging from 3 (worst) to 21 (best). Each item on the LCQ-acute assesses symptoms or the impact of symptoms on HRQoL in the last 24 hours using a 7-point Likert scale ranging from 1 to 7. Higher scores indicate better HRQoL. As per the Statistical Analysis Plan, each domain and total LCQ score change from baseline were analyzed without the treatment by dose interaction. Baseline summaries were evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Days 0 and 22 (Baseline)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1 - Gefapixant | Cohort 1 - Placebo | Cohort 2 - Gefapixant | Cohort 2 - Placebo
Number analyzed (Participants) | 28 | 28 | 30 | 29
Score on a scale
  Psychological Domain Score | 3.8 (1.21) | 4.1 (1.45) | 3.9 (1.57) | 4.1 (1.56)
  Physical Domain Score | 4.4 (0.99) | 4.7 (1.06) | 4.8 (1.19) | 5.0 (1.00)
  Social Domain Score | 4.2 (1.22) | 4.3 (1.21) | 3.9 (1.57) | 4.2 (1.57)
  Total Acute Leicester Score | 12.3 (3.13) | 13.1 (3.41) | 12.6 (4.04) | 13.3 (3.81)

24. Other Pre Specified Outcome: Baseline (Predose) for Cough Visual Analogue Scale (VAS) for Cohort 1 and Cohort 2
Description: Cough VAS: scored from 0 to 100 using a 10 mm visual analogue scale with 0 (no cough) and 100 (most severe cough) mm. Baseline cough VAS is defined as average of screening and baseline cough VAS. Baseline measurements were not available by individual arm because baseline cough frequencies were measured before participants received the first dose of study drug. Baseline summaries were evaluated based on the participant's randomized group (gefapixant or placebo).
Time Frame: Screening, Days 0 and 22 (Baseline)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Cohort 2 - Placebo: Placebo tablet administered by BID daily for 4 days each.
Arm/Group | Cohort 1 - Gefapixant | Cohort 1 - Placebo | Cohort 2 - Gefapixant | Cohort 2 - Placebo
Number analyzed (Participants) | 28 | 28 | 30 | 29
Score on a scale | 58.4 (18.66) | 52.2 (19.21) | 54.5 (24.26) | 57.2 (23.71)

ADVERSE EVENTS:
Time Frame: Adverse event data collection is up to 11 weeks All-cause mortality is up to 22 weeks
Description: Analysis population consisted of all randomized participants who received at least 1 dose of study drug
Groups:
- Cohort 1: Gefapixant 50 mg: Gefapixant 50 mg tablet administered by mouth twice daily (BID) for 4 days.
- Cohort 1: Gefapixant 100 mg: Gefapixant 100 mg tablet administered by mouth BID or 4 days.
- Cohort 1: Gefapixant 200 mg: Gefapixant 200 mg tablet administered by mouth BID for 4 days.
- Cohort 1 - Placebo; Cohort 2- Placebo: Placebo tablet administered by mouth BID for 4 days each.
Arm/Group | Cohort 1: Gefapixant 50 mg | Cohort 1: Gefapixant 100 mg | Cohort 1 - Gefapixant 150 mg | Cohort 1: Gefapixant 200 mg | Cohort 1 - Placebo | Cohort 2 - Gefapixant 7.5 mg | Cohort 2 - Gefapixant 15 mg | Cohort 2 - Gefapixant 30 mg | Cohort 2 - Gefapixant 50 mg | Cohort 2- Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/26 | 0/26 | 0/28 | 0/30 | 0/30 | 0/30 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/28 | 0/26 | 0/26 | 1/28 | 0/30 | 0/30 | 0/30 | 1/30 | 0/29
Other Adverse Events (participants affected / at risk) | 17/28 | 8/28 | 4/26 | 6/26 | 4/28 | 6/30 | 1/30 | 13/30 | 9/30 | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Gefapixant 50 mg (N=28) | Cohort 1: Gefapixant 100 mg (N=28) | Cohort 1 - Gefapixant 150 mg (N=26) | Cohort 1: Gefapixant 200 mg (N=26) | Cohort 1 - Placebo (N=28) | Cohort 2 - Gefapixant 7.5 mg (N=30) | Cohort 2 - Gefapixant 15 mg (N=30) | Cohort 2 - Gefapixant 30 mg (N=30) | Cohort 2 - Gefapixant 50 mg (N=30) | Cohort 2- Placebo (N=29)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Gefapixant 50 mg (N=28) | Cohort 1: Gefapixant 100 mg (N=28) | Cohort 1 - Gefapixant 150 mg (N=26) | Cohort 1: Gefapixant 200 mg (N=26) | Cohort 1 - Placebo (N=28) | Cohort 2 - Gefapixant 7.5 mg (N=30) | Cohort 2 - Gefapixant 15 mg (N=30) | Cohort 2 - Gefapixant 30 mg (N=30) | Cohort 2 - Gefapixant 50 mg (N=30) | Cohort 2- Placebo (N=29)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 13 (13) | 6 (6) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 12 (12) | 4 (4) | 0 (0)
Hypogeusia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No data collected as part of this study will be utilized in any written work, including publications, without the written consent of sponsor.